CLINICAL TRIAL: NCT02450097
Title: Metabolic and Hormonal Effects of 5:2 Intermittent Fasting in Patients With Type 2 Diabetes and Subjects With Adiposity
Brief Title: Metabolic and Hormonal Effects of 5:2 Intermittent Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Kerstin Brismar, M.D/Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Dnr2013/1618-31/3
Record Dates: First submitted 2014-03-24; First posted 2015-05-21 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Obesity; Diabetes Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Other): Intermittent Caloric restriction in 3 Groups:
  I- 40 patients with diabetes type 2 BMI 25.1-37 II- 40 non diabetic over weight subjects with BMI 25.1-37 III- 20 non diabetic subject with BMI 23.1 - 25 and visceral fat
  Interventions: Other: Caloric restriction

INTERVENTIONS:
Other: Caloric restriction

SUMMARY:
The aim of the present study is to investigate in subjects with and without type 2 diabetes the effect of calorie restriction (CR) according to the 5:2 method for 6 months (every week two days caloric fasting with 500 calories for women and 600 calories for men and five days of normal caloric intake) on risk markers for cardiovascular disease and certain cancers (hyperinsulinemia, insulin resistance, IGF-1, IGFBP-1, IGFBP-2, glucose, HbA1c, blood lipids, markers of inflammation and oxidative stress) and on peptides regulating glucose metabolism and appetite as well as the effect on blood pressure, body composition, waist- and hip- circumference. DNA will also be analysed at the start and after 6 months to investigate any epigenetic effects.

After completed study there will be a follow up after additional 6 months.

DETAILED DESCRIPTION:
Background: It is well known that the majority of the population in the western world eats too much calories in relation to physical activity. This results in increased body weight, insulin resistance and premature age-related diseases such as diabetes, hypertension, cardiovascular disease, even dementia and certain types of cancer like colon cancer and breast cancer.

Several studies have shown that calorie restriction (CR) reduces the risk for cardiovascular disease, diabetes and Alzheimer's disease. Animal studies have shown that CR reduces insulin like growth factor-1 (IGF-1) levels, cancer incidence and prolong lifespan. Chronic every day CR decreases blood lipids and glucose, blood pressure, insulin resistance and inflammatory markers. It has been shown to reduce incidence of atherosclerosis directly correlated to the CR and not to weight reduction. However, only few studies have investigated the effect of periodic CR in healthy subjects with adiposity and in patients with type 2 diabetes. Moreover, no studies to our knowledge have studied if there is any gender differences in the metabolic response to periodic CR or if the response is dependent on the degree of adiposity and metabolic disturbance. Since it for many people is very difficult to every day reduce caloric intake , the new method to reduce it to 25% of the normal intake during two days a week is of a great interest to study regarding the metabolic and hormonal effects in men and women.

Questions to be answered; Do women and men respond differently to this diet and do subjects with type 2 diabetes respond differently to those without diabetes. How many subjects can continue to follow this new diet during the 6 months study and during further 6 months follow up?

Primary end points: Change from baseline in fasting serum insulin, C-peptide and insulin like factor binding protein-1 (IGFBP-1) in 6 months.

Secondary end points: Changes in body composition including body fat percentage, blood pressure, blood lipids, blood glucose, markers of inflammation, oxidative stress and hormones regulating appetite, and changes in wellbeing, diet habits and physical activity.

Material/Subjects: 100 subjects will be recruited via media and from outpatient clinics for diabetes care at Karolinska University Hospital and Sophiahemmet Hospital in Stockholm, Sweden.

Method: The subjects who have given informed consent will get a questionnaire regarding well-being, physical activity, life style, family history of diabetes, obesity, hypertension, cardiovascular disease, cancer and of dementia, previous medical and weight history and drugs used. The subjects will be examined by a doctor at a screening visit and blood and urine samples will be taken. Waist and hip circumference, blood pressure and pulse at sitting position after 10 minutes rest, estimation of the body composition, percent body fat and free fat mass (muscle mass) will be registered. The subjects will also respond to a questionnaire regarding diet habits and a meal diary during three ordinary days. A group of 10 to 15 subjects will be informed at a meeting with the doctors, nurses and dietitian about the diet (given 25 examples) during the 2 days of calorie restriction and recommended diet (Mediterranean or Nordic diet) during the other 5 days in the week. The subjects will respond to questions regarding hunger, fullness and satiety during the 2 days of calorie restriction (500 for women and 600 for men) and register which of 25 possible given meals they select during the calorie restriction days every week for 26 weeks. After 6 weeks there will be a follow up with new blood and urine tests, wellbeing questionnaires and after 3 and 6 months new blood and urine test, physical examination, questionnaires regarding physical activity, wellbeing, and diet habits and meal diary during 3 days. After completed study there will be a follow up after additional 6 months when participant are free to choose too continue with CR or not.

At all visits blood pressure, pulse; waist and hip circumference and body composition will be registered. The blood and urine samples will be taken in the morning after an overnight fast and after a day of normal diet. The blood and urine samples will be stored in a local human sample bank at the hospital for later analysis after the study is closed.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years of age.
* Subjects without diabetes with BMI 23-37.
* Patients with Type 2 diabetes and diabetes duration between 0.5-12 years and BMI 25-37

Exclusion criteria:

* BMI below 23
* Waist circumference 80 cm or less for women and 94 cm or less than for men.
* Total fat percent of body weight less than 23%.
* Treatment with insulin and sulfonylurea drugs.
* Chronic kidneys disease (CKD) stage 4 and 5 (eGFR <30 ml/min).
* Pregnancy and breast-feed.
* Active athletes.
* History of eating disorder.
* Participation in another ongoing study.
* If participant is not eligible to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fasting serum insulin in 6 months. | 6 months
  Serum insulin will be measured using a radioimmunoassay (RIA; Pharmacia insulin RIA 100, Pharmacia Diagnostics, Uppsala, Sweden).

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Brismar, Professor, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden